CLINICAL TRIAL: NCT03008070
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter, Dose-range, Proof-of-concept, 24-week Treatment Study of IVA337 in Adult Subjects With Nonalcoholic Steatohepatitis (NASH)
Brief Title: Phase 2b Study in NASH to Assess IVA337
Acronym: NATIVE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Inventiva Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IVA_01_337_HNAS_16_002; 2016-001979-70 (EudraCT Number)
Record Dates: First submitted 2016-12-22; First posted 2017-01-02 (Estimated); Results first posted 2021-04-12 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Non-Alcoholic Steatohepatitis (NASH)
Keywords: Non-Alcoholic Steatohepatitis; NASH; peroxisome proliferator-activated receptor (PPAR); Liver Diseases; Fibrosis; Fatty Liver; Non-alcoholic Fatty Liver Disease; Digestive System Diseases; IVA337
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Liver Diseases; Fibrosis; Fatty Liver; Digestive System Diseases | interventions — lanifibranor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- IVA337 1200mg (Experimental): IVA337 400mg, once a day (Quaque Die, QD) with food
  Interventions: Drug: IVA337
- IVA337 800mg (Experimental): IVA337 400mg, once a day (Quaque Die, QD) with food
  Interventions: Drug: IVA337
- Placebo (Placebo Comparator): Placebo to match, once a day (Quaque Die, QD) with food
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: IVA337 — 1200mg
  Arms: IVA337 1200mg
Drug: IVA337 — 800mg
  Arms: IVA337 800mg
Drug: Placebo — Placebo to match
  Arms: Placebo

SUMMARY:
Non-alcoholic steatohepatitis, abbreviated as NASH, is a chronic liver disease that may progress to cirrhosis. The disease is mostly associated with obesity and type 2 diabetes mellitus, or insulin resistance and is very common. However, Treatment of NASH is a significant unmet clinical need.

IVA337 (lanifibranor) is a next generation pan-PPAR (peroxisome proliferator-activated receptors) agonist addressing the pathophysiology of NASH : metabolic, inflammatory and fibrotic.

The purpose of this research is to evaluate the efficacy and the safety of two doses of IVA337 (800mg, 1200 mg) per day for 24 weeks versus placebo in adult NASH patients with liver steatosis and moderate to severe necroinflammation without cirrhosis.

DETAILED DESCRIPTION:
Randomized (stratified on diabetes), placebo-controlled, double-blind, parallel-assignment, dose-range multicenter study

There are 3 parallel treatment groups: placebo, IVA337 800mg once a day (Quaque Die, QD) and IVA337 1200mg QD (identical tablets of 400mg IVA337 or placebo). Both, patient and investigator are blinded.

For each patient, the study duration will be an overall of 6 to 8 months (with a 10-day to 4-week selection period, a 24-week treatment period and a 4-week follow-up period).

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects, age ≥18 years.
* NASH histological diagnosis according to the currently accepted definition of both EASL and AASLD, requiring the combined presence of steatosis (any degree ≥ 5%) + lobular inflammation of any degree + liver cell ballooning of any amount, on a liver biopsy performed ≤ 6 months before screening in the study or at screening and confirmed by central reading during the screening period and

  * SAF Activity score of 3 or 4 (>2)
  * SAF Steatosis score ≥ 1
  * SAF Fibrosis score < 4
* Subject agrees to have a liver biopsy performed after 24 weeks of treatment.
* Compensated liver disease
* No other causes of chronic liver disease (autoimmune, primary biliary cholangitis, Hepatitis B virus (HBV), hepatitis C virus (HCV), Wilson's, α-1-antitrypsin deficiency, hemochromatosis, etc…).
* If applicable, have a stable type 2 diabetes, defined as HbA1c ≤ 8.5% and fasting glycemia <10 mmol/L, no changes in medication in the previous 6 months, and no new symptoms associated with decompensated diabetes in the previous 3 months.
* Have a stable weight since the liver biopsy was performed defined by no more than a 5 % loss of initial body weight.
* Negative pregnancy test or post-menopausal. Women with childbearing potential (i.e. fertile, following menarche and until becoming post-menopausal unless permanently sterile) must be using a highly effective method of contraception (i.e. combined (estrogen and progestogen containing) hormonal/ progestogen-only hormonal contraception associated with inhibition of ovulation, intrauterine device, intrauterine hormone-releasing system, bilateral tubal occlusion, vasectomised partner). The contraceptive method will have to be followed for at least one menstruation cycle after the end of the study
* Subjects having given her/his written informed consent.

Exclusion Criteria:

* Evidence of another form of liver disease.
* History of sustained excess alcohol ingestion: daily alcohol consumption > 30 g/day (3 drinks per day) for males and > 20 g/day (2 drinks per day) for females.
* Unstable metabolic condition: Weight change > 5kg in the last three months, diabetes with poor glycemic control (HbA1c > 8.5%), introduction of an antidiabetic or of an anti-obesity drug/malabsorptive or restrictive bariatric (weight loss) surgery in the past 6 months prior to screening.
* History of gastrointestinal malabsorptive bariatric surgery within less than 5 years or ingestion of drugs known to produce hepatic steatosis including corticosteroids, high-dose estrogens, methotrexate, tetracycline or amiodarone in the previous 6 months.
* Significant systemic or major illnesses other than liver disease, including congestive heart failure (class C and D of the American Heart Association , AHA), unstable coronary artery disease, cerebrovascular disease, pulmonary disease, renal failure, organ transplantation, serious psychiatric disease, malignancy that, in the opinion of the investigator, would preclude treatment with IVA337 and/or adequate follow up.
* HB antigen >0, HCV Polymerase chain reaction (PCR) tests >0 (patients with a history of HCV infection can be included if HCV PCR is negative since more than 3 years), HIV infection.
* Pregnancy/lactation or inability to adhere to adequate contraception in women of child-bearing potential.
* Active malignancy except cutaneous basocellular carcinoma.
* Any other condition which, in the opinion of the investigator would impede competence or compliance or possibly hinder completion of the study.
* Body mass index (BMI) >45 kg/m2.
* Type 1 diabetes and type 2 diabetic patient on insulin.
* Diabetic ketoacidosis
* Fasting Triglycerides > 300 mg/dL.
* Hemostasis disorders or current treatment with anticoagulants.
* Contra-indication to liver biopsy.
* History of, or current cardiac dysrhythmias and/or a history of cardiovascular disease event, including myocardial infarction, except patients with only well controlled hypertension. Any clinically significant ECG abnormality reported by central ECG reading.
* Participation in any other clinical study within the previous 3 months.
* Have a known hypersensitivity to any of the ingredients or excipients of the Investigational medicinal product (IMP)
* Be possibly dependent on the Investigator or the sponsor (e.g., including, but not limited to, affiliated employee).
* Creatine phosphokinase (CPK)>5 x ULN
* Osteopenia or any other well documented Bone disease. Patient without well documented osteopenia treated with vitamin D and/or Calcium based supplements for preventive reasons can be included.

(The criteria below are applicable only for patients who will undergo a MRI/LMS in selected centers)

* Claustrophobia to a degree that prevents tolerance of MRI scanning procedure. Sedation is permitted at discretion of investigator.
* Metallic implant of any sort that prevents MRI examination including, but not limited to: aneurysm clips, metallic foreign body, vascular grafts or cardiac implants, neural stimulator, metallic contraceptive device, tattoo, body piercing that cannot be removed, cochlear implant; or any other contraindication to MRI examination.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 247 (Actual)
Dates: Start 2017-02-07 (Actual); Primary Completion 2020-02-20 (Actual); Study Completion 2020-03-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sven FRANCQUE, MD, PhD, Principal Investigator — Division of Gastroenterology and Hepatology, Antwerp University Hospital, Wilrijkstraat 10, B-2650 Edegem, Belgium
Locations (85):
- United States (14):
  - North Alabama GI Research Center, Madison, Alabama
  - ACTRI, La Jolla, California
  - National Research Institute, Los Angeles, California
  - Palmetto Research, LLC, Hialeah, Florida
  - Florida Digestive Health Specialists, LLP, Lakewood Rch, Florida
  - Northeast GI Research Division, Concord, Massachusetts
  - Duke University Medical Center, Durham, North Carolina
  - Carolina's Center for Liver Disease/CHG, Huntersville, North Carolina
  - Jefferson University hospital, Philadelphia, Pennsylvania
  - Digestive Health Research, LLC, Hermitage, Tennessee
  - The Texas Liver Institute, San Antonio, Texas
  - Digestive Health Research, LLC, San Antonio, Texas
  - University of Virginia Health System, Charlottesville, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
- Australia (5):
  - Flinders Medical Centre Department of Hepatology, Bedford Park
  - Monash Medical Centre, Clayton
  - Lyell McEwin Hospital & The University of Adelaide, Elizabeth Vale
  - Royal Brisbane and Women's Hospital, Herston
  - Fiona Stanley Hospital, Murdoch
- Medical University Vienna, Vienna, Austria
- Belgium (5):
  - Hopital Erasme, Brussels
  - Clinique Universitaire Saint-luc, Brussels
  - Antwerp University Hospital, Edegem
  - Ziekenhuis Oost Limburg, Genk
  - UZ Gent, Ghent
- Bulgaria (7):
  - "DCC Alexandrovska", EOOD, Sofia
  - Acibadem City Clinic Tokuda Hospital, Sofia
  - Acibadem City Clinic University Hospital EOOD, Sofia
  - MHAT "Sveta Anna" Sofia, Sofia
  - Military Medical Academy - MHAT, Sofia
  - UMHAT "Sv. Ivan Rilski", Sofia
  - UMHAT "Tsaritsa Yoanna-ISUL", Sofia
- Canada (7):
  - University of Calgary, Calgary
  - The Bailey Health Clinic, Edmonton
  - CISSS de la Montérégie Centre, Greenfield Park
  - University of Western Ontario, London Health Sciences Centre, London
  - McGill University Health Centre (MUHC), Montreal
  - Medpharmgene, Inc, Montreal
  - LAIR Centre, Vancouver
- Czechia (3):
  - Researchsite S.R.O., Pilsen
  - Klin Med S.R.O., Prague
  - Institut klinické a experimentální medicíny, IKEM, Prague
- France (14):
  - CHU Angers, Angers
  - CHRU Besançon, Besançon
  - Centre Hospitalier de Bordeaux, Bordeaux
  - CHU Henri Mondor, Créteil
  - CHU de Grenoble, Grenoble
  - Hôpital de La Croix Rousse, Lyon
  - Centre Hospitalier Régional Universitaire de Montpellier, Montpellier
  - CHU de Nice, Nice
  - Hôpital Saint Antoine, Paris
  - Hôpital La Pitié Salpétrière, Paris
  - Hôpital Beaujon, Paris
  - Centre Hospitalier Universitaire de Rennes, Rennes
  - Hôpital de Hautepierre, Strasbourg
  - Hôpital Purpan - Centre Hospitalier Universitaire (CHU) de Toulouse, Toulouse
- Germany (6):
  - RWTH University Hospital, Aachen
  - Innere Medizin II - Universitätsklinik Freiburg, Freiburg im Breisgau
  - Medizinischen Klinik IV, Heidelberg
  - Universitätsmedizin Mainz, I. Med. Klinik, Mainz
  - Universitätsklinikum Münster, Münster
  - University Hospital Würzburg, Würzburg
- Italy (6):
  - Ospedali Riuniti di Ancona-Università Politecnica delle Marche, Ancona
  - Granda Ospedale Maggiore Policlinico - Università di Milano, Milan
  - Pol. Giaccone, Palermo
  - Fondazione Policlinico Agostino Gemelli, Roma
  - Poliambulatorio Giovanni Paolo II, San Giovanni Rotondo
  - A.O. Città della Salute e della Scienza di Torino, Torino
- CAP Research, Quatre Bornes, Mauritius
- Poland (4):
  - Oddzial Gastroenterologii Hepatologii UCK, Katowice
  - Katedra i Klinika Chorób Zakaźnych i Hepatologii Uniwersytetu Medycznego w Łodzi, Lodz
  - Klinika Chorób Zakaźnych, Lublin
  - Centrum Badan Klinicznych, Wroclaw
- Slovenia (2):
  - General hospital Celje, Celje
  - General Hospital Murska Sobota, Murska Sobota
- Spain (5):
  - Vall d'Hebron Hospital, Barcelona
  - Hospital Puerta de Hierro MAJADAHONDA, Madrid
  - Virgen de la Victoria University Hospital, Málaga
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Hospital Virgen del Rocío, Seville
- Switzerland (2):
  - Universitätsklinik für Viszerale Chirurgie und Medizin, Bern
  - Epatocentro Ticino, Lugano
- United Kingdom (3):
  - Kings College Hospital NHS Foundation Trust, London
  - Freeman Hospital, Newcastle University, Newcastle
  - Nottingham University Hospitals NHS Trust, Nottingham

REFERENCES:
- [Derived] Boursier J, Herve H, Roux M, Abdelmalek MF, Francque SM, Broqua P, Junien JL, Abitbol JL, Huot-Marchand P, Dzen L, Cooreman MP, Patel S. Biomarkers of Histological Response in Lanifibranor-treated Patients With Metabolic Dysfunction-associated Steatohepatitis. Clin Gastroenterol Hepatol. 2025 Dec;23(13):2499-2508.e8. doi: 10.1016/j.cgh.2024.12.039. Epub 2025 Mar 17. PMID 40107637
- [Derived] Cooreman MP, Butler J, Giugliano RP, Zannad F, Dzen L, Huot-Marchand P, Baudin M, Beard DR, Junien JL, Broqua P, Abdelmalek MF, Francque SM. The pan-PPAR agonist lanifibranor improves cardiometabolic health in patients with metabolic dysfunction-associated steatohepatitis. Nat Commun. 2024 May 10;15(1):3962. doi: 10.1038/s41467-024-47919-9. PMID 38730247
- [Derived] Francque SM, Bedossa P, Ratziu V, Anstee QM, Bugianesi E, Sanyal AJ, Loomba R, Harrison SA, Balabanska R, Mateva L, Lanthier N, Alkhouri N, Moreno C, Schattenberg JM, Stefanova-Petrova D, Vonghia L, Rouzier R, Guillaume M, Hodge A, Romero-Gomez M, Huot-Marchand P, Baudin M, Richard MP, Abitbol JL, Broqua P, Junien JL, Abdelmalek MF; NATIVE Study Group. A Randomized, Controlled Trial of the Pan-PPAR Agonist Lanifibranor in NASH. N Engl J Med. 2021 Oct 21;385(17):1547-1558. doi: 10.1056/NEJMoa2036205. PMID 34670042
- [Derived] Sven M F, Pierre B, Manal F A, Quentin M A, Elisabetta B, Vlad R, Philippe HM, Bruno S, Jean-Louis J, Pierre B, Jean-Louis A. A randomised, double-blind, placebo-controlled, multi-centre, dose-range, proof-of-concept, 24-week treatment study of lanifibranor in adult subjects with non-alcoholic steatohepatitis: Design of the NATIVE study. Contemp Clin Trials. 2020 Nov;98:106170. doi: 10.1016/j.cct.2020.106170. Epub 2020 Oct 8. PMID 33038502

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment of patients started in February 2017, and last patient was recruited on March 2019. A total of 868 patients were screened for the study.
Pre-assignment Details: Patients were invited to participate into the study by their referent doctor according to the patient's medical records. Patients had to fulfil all the inclusion and none of the exclusion criteria to be eligible.
  A total of 247 patients were randomised, and 621 were not randomised.Main reason for non randomization was inclusion/exclusion criteria not met (470 - 76%).
Groups:
- Lanifibranor 1200mg: Lanifibranor 400mg, once a day (Quaque Die, QD) with food
  Lanifibranor: 1200mg
- Lanifibranor 800mg: Lanifibranor 400mg, once a day (Quaque Die, QD) with food
  Lanifibranor: 800mg
Period: Overall Study
Arm/Group | Lanifibranor 1200mg | Lanifibranor 800mg | Placebo
Started | 83 | 83 | 81
Completed | 77 | 77 | 74
Not Completed | 6 | 6 | 7
Not completed — Adverse Event | 3 | 3 | 3
Not completed — Lost to Follow-up | 1 | 1 | 0
Not completed — Non compliance | 0 | 1 | 1
Not completed — Withdrawal by patient and adverse event non fatal | 0 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 1
Not completed — Use of prohibited drug | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IVA337 1200mg | IVA337 800mg | Placebo | Total
Number analyzed (Participants) | 83 | 83 | 81 | 247
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 67 | 69 | 63 | 199
  >=65 years | 16 | 14 | 18 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.2 (13.8) | 55 (10.4) | 53.4 (13.1) | 53.6 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 54 | 41 | 144
  Male | 34 | 29 | 40 | 103
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 2 | 2
  Asian | 2 | 1 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Black or African American | 3 | 1 | 3 | 7
  White | 78 | 80 | 74 | 232
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 13 | 11 | 12 | 36
  Czechia | 3 | 2 | 3 | 8
  United Kingdom | 3 | 2 | 2 | 7
  Mauritius | 2 | 3 | 2 | 7
  Switzerland | 0 | 3 | 1 | 4
  Spain | 3 | 4 | 5 | 12
  Canada | 3 | 1 | 4 | 8
  Austria | 0 | 1 | 0 | 1
  Belgium | 10 | 11 | 11 | 32
  Poland | 1 | 2 | 3 | 6
  Italy | 3 | 1 | 1 | 5
  Slovenia | 0 | 1 | 0 | 1
  Australia | 3 | 7 | 3 | 13
  Bulgaria | 17 | 16 | 22 | 55
  France | 15 | 15 | 9 | 39
  Germany | 7 | 3 | 3 | 13

OUTCOME MEASURES:

1. Primary Outcome: SAF Activity Score (SAF-A) Decrease of at Least 2 Points With no Worsening of the CRN Fibrosis Score (CRN-F)
Description: SAF-A is the activity part of the Steatosis Activity Fibrosis [SAF] histological score, calculated as the sum of lobular inflamation score and balloning score.
  No worsening of fibrosis means that the CRN fibrosis score (CRN-F) remains stable or decreases.
Time Frame: 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | IVA337 1200mg | IVA337 800mg | Placebo
Number analyzed (Participants) | 83 | 83 | 81
Participants
  Yes | 41 | 34 | 22
  No | 42 | 49 | 59
Statistical Analysis 1: Comparison: IVA337 800mg vs Placebo; The primary endpoint was a binary outcome (Yes/No). Responders rates were compared between the placebo and lanifibranor 800 mg at the end of the treatment period (week 24) using a Cochran Mantel Haenzel test stratified on diabetic status at baseline (that was the stratified factors in the randomisation). The CMH risk ratio is used to estimate the effect size. Patients with missing data are considered as non-responders; Test type: Superiority; p = 0.061, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 1.52, 95% CI 2-sided [0.98 to 2.12]
Statistical Analysis 2: Comparison: IVA337 1200mg vs Placebo; The primary endpoint was a binary outcome (Yes/No). Responders rates were compared between the placebo and lanifibranor 1200 mg at the end of the treatment period (week 24) using a Cochran Mantel Haenzel test stratified on diabetic status at baseline (that was the stratified factors in the randomisation). The CMH risk ratio is used to estimate the effect size. Patients with missing data are considered as non-responders; Test type: Superiority; p = 0.004, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 1.82, 95% CI 2-sided [1.24 to 2.4]

2. Secondary Outcome: NASH Improvement
Description: NASH improvement is defined as a decrease of at least 2 points in NAS score (sum of CRN Steatosis, Inflammation and Ballooning scores) without worsening of CRN Fibrosis score.
Time Frame: 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | IVA337 1200mg | IVA337 800mg | Placebo
Number analyzed (Participants) | 83 | 83 | 81
Participants
  Yes | 53 | 43 | 26
  No | 30 | 40 | 55

3. Secondary Outcome: NASH Resolution and no Worsening of Fibrosis
Description: Resolution of NASH is defined as a CRN Inflammation score equal to 0 or 1, and a CRN Ballooning score equal to 0. No worsening of fibrosis means that the CRN fibrosis score remains stable or decreases.
Time Frame: 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | IVA337 1200mg | IVA337 800mg | Placebo
Number analyzed (Participants) | 83 | 83 | 81
Participants
  Yes | 37 | 27 | 15
  No | 46 | 56 | 66

4. Secondary Outcome: Improvement of Fibrosis by at Least 1 Stage and no Worsening of NASH
Description: Improvement of fibrosis is defined as a decrease of at least one stage in CRN Fibrosis score. No worsening of NASH is defined as no increase of CRN Steatosis score, no increase of CRN Inflammation score ans no increase of CRN Ballooning score.
Time Frame: 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | IVA337 1200mg | IVA337 800mg | Placebo
Number analyzed (Participants) | 83 | 83 | 81
Participants
  Yes | 35 | 23 | 19
  No | 48 | 60 | 62

5. Secondary Outcome: Activity (SAF-A) Improvement
Description: SAF-A is the activity part of the Steatosis Activity Fibrosis [SAF] histological score, calculated as the sum of lobular inflamation score and balloning score. Improvement of SAF-A is defined as a decrease of at least 1 point.
Time Frame: 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | IVA337 1200mg | IVA337 800mg | Placebo
Number analyzed (Participants) | 83 | 83 | 81
Participants
  Yes | 62 | 54 | 40
  No | 21 | 29 | 41

6. Secondary Outcome: Steatosis (CRN-S) Improvement
Description: Improvement of CRN Steatosis score (CRN-S) is defined as a decrease of at least 1 point.
Time Frame: 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | IVA337 1200mg | IVA337 800mg | Placebo
Number analyzed (Participants) | 83 | 83 | 81
Participants
  Yes | 54 | 46 | 21
  No | 29 | 37 | 60

7. Secondary Outcome: Lobular Inflammation (CRN-I) Improvement
Description: Improvement of CRN Lobular inflammation score (CRN-I) is defined as a decrease of at least 1 point.
Time Frame: 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | IVA337 1200mg | IVA337 800mg | Placebo
Number analyzed (Participants) | 83 | 83 | 81
Participants
  Yes | 43 | 34 | 30
  No | 40 | 49 | 51

8. Secondary Outcome: Hepatocyte Balooning (CRN-B) Improvement
Description: Improvement of CRN Ballooning (CRN-B) is defined as a decrease of at least 1 point.
Time Frame: 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | IVA337 1200mg | IVA337 800mg | Placebo
Number analyzed (Participants) | 83 | 83 | 81
Participants
  Yes | 60 | 54 | 37
  No | 23 | 29 | 44

9. Secondary Outcome: Fibrosis (CRN-F) Improvement
Description: Improvement of CRN Fibrosis score (CRN-F) is defined as a decrease of at least 1 point.
Time Frame: 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | IVA337 1200mg | IVA337 800mg | Placebo
Number analyzed (Participants) | 83 | 83 | 81
Participants
  Yes | 36 | 28 | 22
  No | 47 | 55 | 59

10. Secondary Outcome: Modified ISHAK Fibrosis (ISHAK-F) Improvement
Description: Improvement of Modified ISHAK Fibrosis (ISHAK-F) is defined as a decrease of at least 1 point.
Time Frame: 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | IVA337 1200mg | IVA337 800mg | Placebo
Number analyzed (Participants) | 83 | 83 | 81
Participants
  Yes | 41 | 32 | 25
  No | 42 | 51 | 56

11. Secondary Outcome: Absolute Change in ALT
Description: Absolute change is defined as Week 24 value - baseline value. Baseline value was defined as the last available non-missing data before or equal to the treatment start.
Time Frame: 24 weeks
Measure: Mean (Standard Error); unit: U/L
Arm/Group | IVA337 1200mg | IVA337 800mg | Placebo
Number analyzed (Participants) | 74 | 72 | 72
U/L | -24.54 (3.82) | -26.08 (3.85) | -1.4 (3.88)

12. Secondary Outcome: Absolute Change in AST
Description: as for outcome 11
Time Frame: 24 weeks
Measure: Mean (Standard Error); unit: U/L
Arm/Group | IVA337 1200mg | IVA337 800mg | Placebo
Number analyzed (Participants) | 74 | 72 | 72
U/L | -12.04 (3.17) | -15.11 (3.2) | -0.08 (3.22)

13. Secondary Outcome: Absolute Change in GGT
Description: as for outcome 11
Time Frame: 24 weeks
Measure: Mean (Standard Error); unit: U/L
Arm/Group | IVA337 1200mg | IVA337 800mg | Placebo
Number analyzed (Participants) | 74 | 72 | 73
U/L | -27.87 (5.57) | -43.38 (5.61) | 4.41 (5.65)

14. Secondary Outcome: Absolute Change in Fibrinogen
Description: as for outcome 11
Time Frame: 24 weeks
Measure: Mean (Standard Error); unit: g/L
Arm/Group | IVA337 1200mg | IVA337 800mg | Placebo
Number analyzed (Participants) | 73 | 69 | 73
g/L | -0.14 (0.81) | -0.10 (0.61) | 0.02 (0.67)

15. Secondary Outcome: Absolute Change in Hs-CRP
Description: as for outcome 11
Time Frame: 24 weeks
Measure: Mean (Standard Error); unit: mg/L
Arm/Group | IVA337 1200mg | IVA337 800mg | Placebo
Number analyzed (Participants) | 74 | 72 | 72
mg/L | -1.37 (0.46) | -2.05 (0.47) | 0.11 (0.47)

16. Secondary Outcome: Absolute Change in Alpha2 Macroglobulin
Description: as for outcome 11
Time Frame: 24 weeks
Measure: Mean (Standard Error); unit: g/L
Arm/Group | IVA337 1200mg | IVA337 800mg | Placebo
Number analyzed (Participants) | 72 | 68 | 71
g/L | 0.13 (0.38) | 0.15 (0.40) | 0.05 (0.35)

17. Secondary Outcome: Absolute Change in Haptoglobulin
Description: as for outcome 11
Time Frame: 24 weeks
Measure: Mean (Standard Error); unit: g/L
Arm/Group | IVA337 1200mg | IVA337 800mg | Placebo
Number analyzed (Participants) | 74 | 72 | 72
g/L | -0.099 (0.378) | -0.053 (0.256) | 0.074 (0.291)

18. Secondary Outcome: Absolute Change of Fasting Plasma Glucose
Description: Absolute change is defined as Week 24 value - baseline value. Baseline value was defined as the last available non-missing data before or equal to the treatment start. Only fasting values were considered.
Time Frame: 24 weeks
Measure: Mean (Standard Error); unit: mmol/L
Arm/Group | IVA337 1200mg | IVA337 800mg | Placebo
Number analyzed (Participants) | 73 | 71 | 72
mmol/L | -0.6 (0.12) | -0.78 (0.12) | 0.24 (0.12)

19. Secondary Outcome: Absolute Change in Insulin
Description: as for outcome 18
Time Frame: 24 weeks
Measure: Mean (Standard Error); unit: pmol/L
Arm/Group | IVA337 1200mg | IVA337 800mg | Placebo
Number analyzed (Participants) | 65 | 68 | 66
pmol/L | -114.91 (11.75) | -118.66 (11.66) | -35.7 (11.6)

20. Secondary Outcome: Absolute Change in HOMA Index
Description: as for outcome 18
Time Frame: 24 weeks
Measure: Mean (Standard Error); unit: index
Arm/Group | IVA337 1200mg | IVA337 800mg | Placebo
Number analyzed (Participants) | 63 | 64 | 65
index | -5.46 (0.58) | -5.79 (0.58) | -1.47 (0.57)

21. Secondary Outcome: Absolute Change in HbA1c
Description: as for outcome 18
Time Frame: 24 weeks
Measure: Mean (Standard Error); unit: percentage
Arm/Group | IVA337 1200mg | IVA337 800mg | Placebo
Number analyzed (Participants) | 74 | 72 | 72
percentage | -0.41 (0.05) | -0.38 (0.05) | 0.07 (0.05)

22. Secondary Outcome: Absolute Change in Total Cholesterol
Description: as for outcome 18
Time Frame: 24 weeks
Measure: Mean (Standard Error); unit: mmol/L
Arm/Group | IVA337 1200mg | IVA337 800mg | Placebo
Number analyzed (Participants) | 74 | 72 | 73
mmol/L | -0.07 (0.07) | -0.02 (0.08) | 0.01 (0.08)

23. Secondary Outcome: Absolute Change of HDL-Cholesterol
Description: as for outcome 18
Time Frame: 24 weeks
Measure: Mean (Standard Error); unit: mmol/L
Arm/Group | IVA337 1200mg | IVA337 800mg | Placebo
Number analyzed (Participants) | 74 | 71 | 73
mmol/L | 0.11 (0.02) | 0.16 (0.02) | 0.01 (0.02)

24. Secondary Outcome: Absolute Change of LDL-Cholesterol
Description: as for outcome 18
Time Frame: 24 weeks
Measure: Mean (Standard Error); unit: mmol/L
Arm/Group | IVA337 1200mg | IVA337 800mg | Placebo
Number analyzed (Participants) | 73 | 71 | 69
mmol/L | 0.03 (0.07) | 0.03 (0.07) | 0.01 (0.07)

25. Secondary Outcome: Absolute Change in Triglycerides
Description: as for outcome 18
Time Frame: 24 weeks
Measure: Mean (Standard Error); unit: mmol/L
Arm/Group | IVA337 1200mg | IVA337 800mg | Placebo
Number analyzed (Participants) | 74 | 71 | 72
mmol/L | -0.44 (0.09) | -0.49 (0.09) | 0.06 (0.09)

26. Secondary Outcome: Absolute Change in Apo A1
Description: as for outcome 18
Time Frame: 24 weeks
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | IVA337 1200mg | IVA337 800mg | Placebo
Number analyzed (Participants) | 73 | 72 | 72
mg/dL | -4.39 (2.16) | -0.29 (2.19) | 0.03 (2.18)

27. Secondary Outcome: Absolute Change in Adiponectin
Description: as for outcome 18
Time Frame: 24 weeks
Measure: Mean (Standard Error); unit: microgram/mL
Arm/Group | IVA337 1200mg | IVA337 800mg | Placebo
Number analyzed (Participants) | 73 | 66 | 72
microgram/mL | 17.12 (1.44) | 11.95 (1.51) | -0.35 (1.44)

28. Secondary Outcome: Resolution of NASH and Improvement of Fibrosis by at Least 1 Stage
Description: Resolution of NASH is defined as a CRN Inflammation score equel to 0 or 1, and a CRN ballooning score equal to 0. Improvement of firbosis is defined as a decrease of at least one stage in CRN Fibrosis score.
Time Frame: From baseline to Week 24.
Measure: Count of Participants; unit: Participants
Arm/Group | Lanifibranor 1200mg | Lanifibranor 800mg | Placebo
Number analyzed (Participants) | 83 | 83 | 81
Participants
  Yes | 26 | 17 | 6
  No | 57 | 66 | 75

ADVERSE EVENTS:
Time Frame: On or after the first dose of treatment up to 30 days post last dose.
Arm/Group | IVA337 1200mg | IVA337 800mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/83 | 0/83 | 0/81
Serious Adverse Events (participants affected / at risk) | 7/83 | 3/83 | 3/81
Other Adverse Events (participants affected / at risk) | 60/83 | 48/83 | 30/81
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IVA337 1200mg (N=83) | IVA337 800mg (N=83) | Placebo (N=81)
Post procedural haematoma (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumobilia (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Undifferentiated connective tissue disease (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Foot operation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IVA337 1200mg (N=83) | IVA337 800mg (N=83) | Placebo (N=81)
Weight increased (Investigations) | 7 (7) | 8 (8) | 0 (0)
Transaminases increased (Investigations) | 3 (3) | 5 (5) | 1 (1)
Headache (Nervous system disorders) | 7 (7) | 4 (6) | 4 (5)
Dizziness (Nervous system disorders) | 6 (6) | 2 (3) | 3 (3)
Fatigue (General disorders) | 11 (11) | 3 (3) | 8 (8)
Oedema peripheral (General disorders) | 7 (7) | 5 (5) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 10 (11) | 8 (8) | 1 (2)
Nausea (Gastrointestinal disorders) | 7 (7) | 8 (8) | 3 (3)
Constipation (Gastrointestinal disorders) | 5 (5) | 3 (3) | 6 (6)
Viral upper respiratory tract infection (Infections and infestations) | 3 (5) | 3 (4) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-07-09): https://cdn.clinicaltrials.gov/large-docs/70/NCT03008070/Prot_002.pdf
  • Statistical Analysis Plan (2020-05-13): https://cdn.clinicaltrials.gov/large-docs/70/NCT03008070/SAP_003.pdf